CLINICAL TRIAL: NCT00804180
Title: Evaluation of a Group Therapy Intervention for Children and Adolescents With Injection-Related Anxiety and Their Caregivers
Brief Title: Group Therapy Intervention for Children and Adolescents With Injection-Related Anxiety and Their Caregivers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment/participants
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Matt Jandrisevits, Psychologist, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHW 08/137, GC 742
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Anxiety
Keywords: anxiety; injection; needle; pediatric; youth; children; adolescents; cognitive behavioral; behavioral; exposure; group; treatment; chronic illness; adherence
MeSH Terms: conditions — Anxiety Disorders; Behavior; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coping skills intervention (Other): Self-Injection Anxiety Counseling: Evaluation of a group treatment for injection-related anxiety. The intention of the study is to obtain basic evaluation of a clinical treatment offered in a natural clinic setting, and does not include a control group, or procedure for random assignment of participants.
  Interventions: Behavioral: Self-Injection Anxiety Counseling

INTERVENTIONS:
Behavioral: Self-Injection Anxiety Counseling — This 5-session group intervention involves: psychoeducation; physiological treatment of anxiety though the instruction and practice of relaxation techniques; cognitive restructuring for anxiety-reduction; practice physiological and cognitive treatments through in vivo injection procedures; and problem solving strategies to generalize treatment gains.

SUMMARY:
The specific aim of this project is to determine the impact of this group therapy intervention on improving adherence, coping, and functioning among children and adolescents with disease processes requiring injections who experience injection-related anxiety.Hypotheses include:

1. General psychosocial (quality of life) improvements from beginning to post-treatment as well as maintenance of these improvements 2-4 weeks following the termination of treatment for both youth and parents.
2. Reduced injection-related anxiety from baseline to post-treatment as well as maintenance of this improvement 2-4 weeks following the end of treatment for both youth and parents.
3. Reduced anxiety immediately following exposure to feared injection- related stimuli.
4. For participants experiencing poor adherence to medical treatment, improvement in adherence as reported by both parents and youth from baseline to post-treatment as well as maintenance of these improvements 2-4 weeks following the end of treatment.

DETAILED DESCRIPTION:
The proposed intervention protocol is a modification of an existing empirically developed treatment (Self-Injection Anxiety Counseling) for adults with injection related anxiety who rely on self-injection for illness management (Mohr, Cox, & Boudewyn, 2003). Self-Injection Anxiety Counseling (SIAC) was developed to assist psychologists and medical staff in working with patients individually to develop strategies to reduce anxiety and increase an individual's ability to self-inject. This treatment protocol has been found to result in increased self injection in patients who experienced injection anxiety prior to undergoing this treatment (Mohr, Cox, & Merluzzi, 2005). Permission has been obtained from Dr. Mohr to modify this treatment manual to be applied to youth in group setting.

This modified group protocol consists of five group sessions. The goals of the first session include development of a group identity, psychoeducation, and physiological treatment of anxiety though the instruction and practice of relaxation techniques. The second session introduces a cognitive component to anxiety reduction and focuses on unhelpful thoughts and strategies youth and caregivers can use to counteract these thoughts. The third session implements the previously learned physiological and cognitive treatments through in vivo injection practice. A registered nurse skilled in working with youth and caregivers on self-injection will be present and active throughout this session and all infection control procedures will be followed. Problem solving strategies are implemented in the fourth session to reduce any difficulties encountered by participants as they practiced their injection goal throughout the week. The fifth session will occur two weeks after the fourth session. This extra week between sessions allows for additional practice and problem solving related to injection goals. The last session reviews problem solving strategies and celebrates the success of participants.

Relevant outcomes for hypotheses testing will be measured before treatment, after completion of treatment, and at follow-up; one measure of injection-related anxiety will be utilized more frequently throughout the treatment.

ELIGIBILITY:
Inclusion Criteria:

* children/adolescents aged 8-17 years.
* presence of a regular caregiver who can participate in weekly group sessions
* injection-related anxiety resulting in either inadequate compliance with injections or significant distress during injections

Exclusion Criteria:

* severe cognitive impairment
* aggression and/or dangerous behavior in the last six months
* currently at risk of harm to themselves or others
* extreme mood lability
* poorly controlled comorbid psychiatric disorders
* active substance use
* current significant legal involvement
* anxiety that impairs daily functioning beyond injections

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory: (Spielberger, 1983) | intake, post-treatment, follow-up (2-4wks)

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory - Generic Core Scales (PedsQL) - Short Form: (Varni, Seid, & Kurtin, 2001) | intake, post-treatment, follow-up (2-4wks)
Subjective Units of Distress Scale | intake, before/after exposures during group sessions, post-treatment, follow-up (2-4wks)
Parental Report of Child's Injection Adherence Percentage (over period of 10 physician-prescribed injection time points) | intake, post-treatment, follow-up (2-4wks)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Jandrisevits, PhD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States